CLINICAL TRIAL: NCT04815746
Title: Psychosocial Determinants of Health-Related Quality of Life (QOL) and Gastrointestinal (GI) Functional Outcomes During Treatment for Malignancies
Brief Title: QOL and GI Outcomes in Malignancies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We have decided to withdraw this research study due to the receipt of funding for a similar study that aligns more closely with our current research priorities and available resources.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190846
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Psychological Adaptation; Psychological Adjustment; Stress, Emotional
Keywords: Psychosocial Symptom Management; eHealth Intervention
MeSH Terms: conditions — Stress, Psychological | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial Symptom Management Intervention (PSMI) Experimental Condition Arm (Experimental): Participants in this group will receive the Cognitive Behavioral Therapy (CBT)-based skills over a 10-week period.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)-based skills
- Usual Clinical Care Control Arm (Active Comparator): Participants in this group will receive standard education.
  Interventions: Behavioral: Standard Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT)-based skills — The CBT skills target reducing anxiety, (e.g., relaxation), changing negative appraisals (e.g., cognitive restructuring), coping skills training (e.g., enhancing adaptive skills), behavioral activation, interpersonal skills (e.g., communication skills) and building or enhancing social networks. The intervention will be administered online, and each module will last about 1-hour.
  Arms: Psychosocial Symptom Management Intervention (PSMI) Experimental Condition Arm
Behavioral: Standard Education — Patients randomized to standard clinical care will receive standard education based on various resources (e.g., National Cancer Institute) relevant to pancreatic cancer.
  Arms: Usual Clinical Care Control Arm

SUMMARY:
The purpose of this research is to evaluate a new, web-based program among patients with pancreatic cancer aimed at reducing psychosocial stress.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years of age
2. Spanish or English speaker with ability to read one of these languages
3. Diagnosis of pancreatic cancer .
4. Willingness to be assessed at diagnosis, during neoadjuvant chemotherapy (if applicable), preoperatively (if applicable - unless time of diagnosis is preoperative visit), and postoperatively for up to two years following surgery.

Exclusion Criteria:

1. Patients unable to read Spanish or English, as they will be unable to complete surveys.
2. History of previous invasive cancer or treatment with chemotherapy, as they may have a different baseline functional status, quality of life, and gastrointestinal function compared to the normal healthy population, per principal investigator discretion, based on a case-by-case review.
3. Prior inpatient psychiatric treatment for severe mental illness or overt signs of severe psychopathology (e.g., psychosis) within the past six months as these conditions can interfere with adequate participation in assessments, per principal investigator discretion, based on a case-by-case review.
4. Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life as Measured by Perceived Stress Scale | Up to 10 weeks.
  Perceived Stress Scale (Scale of 1-40 with higher scores indicating higher stress)
Health Related Quality of Life as Measured by University of California, Los Angeles (UCLA) Loneliness Scale | Up to 10 weeks.
  UCLA Loneliness Scale (Scale of 20-80 with higher scores indicating higher loneliness)
Health Related Quality of Life as Measured by Interpersonal Support Evaluation List | Up to 10 weeks.
  Interpersonal Support Evaluation List (12 item questionnaire evaluated on a 4-point Likert scale with a higher score indicating higher support).
Health Related Quality of Life as Measured by Functional Assessment of Cancer Therapy General - 7 Item Version (FACT-G7) | Up to 10 weeks.
  FACT-G7 (Scale of 0-28 with higher scores indicating better quality of life)
Health Related Quality of Life as Measured by Functional Assessment of Cancer Therapy (FACT) Hepatobiliary-Pancreatic Symptom Index (FHSI)-18 | Up to 10 weeks.
  FACT FHSI-18 (Scale of 0-72 with lower scores indicating better quality of life)
The Gastrointestinal Symptom Rating Scale (GSRS) | Up to 10 weeks.
  GSRS (Scale of 0-78 with higher scores indicating worse gastrointestinal symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Penedo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No